CLINICAL TRIAL: NCT03960684
Title: Prospective Study of Colorectal Procedures With the Levita Magnetic Surgical System
Brief Title: Study of Colorectal Procedures With the Levita Magnetic Surgical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP006
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Levita Magnetic Surgical System (Experimental): Levita Magnetic Surgical System
  Interventions: Device: Levita Magnetic Surgical System

INTERVENTIONS:
Device: Levita Magnetic Surgical System — Levita Magnetic Surgical System

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Levita Magnetic Surgical System in patients undergoing colorectal procedures.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm, open label study designed to assess the safety and effectiveness of the Levita Magnetic Surgical System in colorectal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject is scheduled to undergo elective colorectal surgery

Exclusion Criteria:

* Significant comorbidities
* Subjects with pacemakers, defibrillators, or other electromedical implants
* Subjects with ferromagnetic implants
* Clinical history of impaired coagulation
* Subject has an anatomical abnormality noted after initiation of index procedure that would prevent device use
* Subject is not likely to comply with the follow-up evaluation schedule
* Subject is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I. Emre Gorgun, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Hospital del Salvador, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levita Magnetic Surgical System
Started | 31
Completed | 30
Not Completed | 1
Not completed — Did not proceed to surgery with MSS | 1

BASELINE CHARACTERISTICS:
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 subject did not proceed with procedure. Data was not analyzed.
  years
    number analyzed (Participants) | 30
    (all) | 63 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject did not proceed with procedure and data was not analyzed.
  Participants
    number analyzed (Participants) | 30
    Female | 15
    Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject did not proceed with procedure. Data was not analyzed.
  Participants
    number analyzed (Participants) | 30
    Hispanic or Latino | 30
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 31

OUTCOME MEASURES:

1. Primary Outcome: Number and Types of Tools Required to Retract the Colon or Peri-colorectal Tissues
Description: Ability to adequately retract the colon, peri-colorectal tissues or adjacent organs to achieve an effective exposure of the target tissue. Adequate retraction is achieved if it is not necessary to replace the Levita Magnetic Surgical System with another instrument to retract these tissues during the procedure.
  Cumulative number of additional tools required across all participants.
Time Frame: During planned colorectal procedure
Measure: Number; unit: Cumulative number of additional tools
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 30
Cumulative number of additional tools | 0

2. Primary Outcome: Device Related Adverse Events
Description: All adverse events will be recorded and allocated as to relatedness to device, procedure or other.
Time Frame: Through 30 days post colorectal procedure/study completion.
Measure: Number; unit: Number of Device Related Adverse Events
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 30
Number of Device Related Adverse Events | 6

ADVERSE EVENTS:
Time Frame: 30 days post-procedure
Arm/Group | Levita Magnetic Surgical System
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levita Magnetic Surgical System (N=30)
Dehiscence Colorectal Anastomosis (Gastrointestinal disorders) | 1 (1)
Pelvic Fluid Collection in Relation to Ileal Pouch (Gastrointestinal disorders) | 1 (1)
Mechanical Ileus Obstruction (Gastrointestinal disorders) | 1 (1)
Clostridium Infection (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levita Magnetic Surgical System (N=30)
Petechias Peritoneal (Gastrointestinal disorders) | 5 (5)
Wound Infection (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03960684/Prot_SAP_000.pdf